CLINICAL TRIAL: NCT05206526
Title: DRagonboat Activity for CAncer RecoverY and Self-efficacy
Brief Title: Dragonboat Activity for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRACARYS
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dragon Boat (Experimental): 12 weeks of training, defined by a precise progressive, structured and supervised program divided into 3 weekly sessions of one hour / one hour and a half preparatory to the Dragon Boat activity.
  Interventions: Behavioral: Dragon Boat
- Control (Active Comparator): 12 weeks of home-based training, without supervision, to perform 3 time per week composed by ten total body exercise.
  Interventions: Behavioral: Home-based Exercise

INTERVENTIONS:
Behavioral: Dragon Boat — 12 weeks of training, defined by a precise progressive, structured and supervised program divided into 3 weekly sessions of one hour / one hour and a half preparatory to the Dragon Boat activity.
  Arms: Dragon Boat
Behavioral: Home-based Exercise — 12 weeks of home-based training composed by 10 exercises.
  Arms: Control

SUMMARY:
The goal of this study is to determine how a structured and supervised physical activity program linked to Dragon Boat practice can improve motivation to participate in physical activity sessions. It is also the purpose of this study to evaluate the improvement in body composition, body image perception and physical function.

For this purpose, a group of women operated on for breast cancer was recruited and divided into two experimental groups: one group participated in a structured program of Dragon Boat while the other followed a home-based program of exercises independently in the home environment.

Anthropometric measures (weight, height, BMI) and arm circumference, data on lifestyle and psychological well-being were evaluated by means of questionnaires. Tests were also performed to assess shoulder strength, aerobic capacity and mobility.

The results of this study will (a) identify the strategies used that make Dragon Boat activity effective in ensuring quality participation in physical activity, (b) define the physiological effects of Dragon Boat activity on physical functionality and (c) correlating objective measures with subjective perceptions thanks to the integration of new body composition analysis techniques (regional BIA) and validated questionnaires on the perception of body image.

ELIGIBILITY:
Inclusion Criteria:

* age 45-70 years
* Body mass index: <18 and <30 kg / m2
* Diagnosis and treatment for breast cancer

Exclusion Criteria:

* Other corneal diseases (cardiovascular, hepatic, respiratory)
* Participation in other structured exercise programs

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Lean body mass | Change from baseline to up to 3 months
  kilograms of muscle mass measure by bioimpendenziometry
cardiovascular fitness | Change from baseline to up to 3 months
  meters walked during the 6 minutes walking test
body appreciation | Change from baseline to up to 3 months
  body image perception measured by the score of the Body Appreciation Scale-2 rated on a 5-point Likert-type scale ranging from Never (receiving a score of 1) to Always (receiving a score of 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moro T, Casolo A, Bordignon V, Sampieri A, Schiavinotto G, Vigo L, Ghisi M, Paoli A, Cerea S. Keep calm and keep rowing: the psychophysical effects of dragon boat program in breast cancer survivors. Support Care Cancer. 2024 Mar 8;32(4):218. doi: 10.1007/s00520-024-08420-7. PMID 38456933